CLINICAL TRIAL: NCT06822660
Title: Dreams or Implicite Memorization Under OFA
Acronym: Dreams
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Other Study IDs: B0762024241010
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Implicite Memorization
Keywords: implicite memorization; opioid free anesthesia; observationnal; monocentric; isolated forearm technique; explicite memorization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Dreams study is an observational study aimed at evaluating the incidence of connected awareness after intubation, intraoperative explicit and implicit memorization, and postoperative well-being in patients receiving general anesthesia without opioids.

Outcomes

The primary objective is the evaluation of the incidence of connected consciousness after induction of general anesthesia without opioids and intubation. The secondary objectives are:

* Implicit and explicit memorization after intubation and during the procedure
* Post-operative well-being Pain in the recovery room and in the room, assessed by VAS;
* Total consumption of analgesics (paracetamol, diclofenac, tramadol): data collected during discharge
* Level of satisfaction, assessed using the EVAN scale
* Duration of hospitalization
* Estimated first mobilization

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic robotic surgery
* ASA score 1 to 3

Exclusion Criteria:

* neurological and psychiatric diseases
* reflect memory disorders
* head trauma
* hearing disorders
* past or current use of medications affecting the central nervous system.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We study patients 18-75 aged undergoing laparoscopic robotic surgery ( prostatectomy, hysterectomy, colectomy) with an ASA status from 1 to 3.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Implicite memorization incidence | From the operating room to one week after surgery
  Through the isolated forearm technique and with the capacity of patients to recognize post operatively sounds that they have listened during the anesthesia, we evaluate the incidence of implicite memorization

SECONDARY OUTCOMES:
explicite memorization | From the operating room to one week after surgery
  Through the modified brice questionnaire, we assess the incidence of explicite memorization

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Saint Pierre, Brussels, Belgium